CLINICAL TRIAL: NCT04896138
Title: A Study of the Natural Progression of Interstitial Lung Disease
Brief Title: University of Virginia Natural History Study
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Imre Noth, MD, Professor, University of Virginia
Other Study IDs: 20937
Record Dates: First submitted 2021-04-26; First posted 2021-05-21 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis; Sarcoidosis; Connective Tissue Diseases; Hypersensitivity Pneumonitis; Idiopathic Interstitial Pneumonias
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis; Sarcoidosis; Connective Tissue Diseases; Alveolitis, Extrinsic Allergic; Idiopathic Interstitial Pneumonias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ILD Cohort: Patients with Interstitial Lung Disease seen at the UVA ILD or Pulmonary Clinic
  Interventions: Other: Interstitial Lung Disease
- Control Cohort: Control group of patients and family members of those with an Interstitial Lung Disease

INTERVENTIONS:
Other: Interstitial Lung Disease — Not applicable - this is not an interventional trial
  Groups: ILD Cohort

SUMMARY:
Data and specimens will be collected longitudinally from patients seen in the UVA Interstitial Lung Disease (ILD) clinic in order to describe the phenotypic expression of various interstitial lung diseases. Samples will also be collected from a control group for comparison purposes.

All data will be entered into a repository for future research purposes or screening for new studies that become available. This data will help identify trends and hopefully lead to a better understanding of the disease progression, treatment options, and outcomes.

DETAILED DESCRIPTION:
Following the clinical course of patients with ILD will allow description of the natural history of these diseases and prospective analysis of the following specific questions:

1. Can surrogate physiological markers of disease progression be used in place of mortality? Mortality of a defined cohort of patients will be developed. The surrogate markers include but are not limited to serial cardiopulmonary exercise testing, pulmonary function testing, 6-minute walk testing, HRCT scanning and echocardiography.
2. Do alternative assessments such as quality of life (QOL) questionnaires provide early prediction of physiological change as measured by the previously described parameters? Periodic QOL questionnaires are regularly conducted in clinic and will be followed
3. Does rate of deterioration as measured by these previously described parameters affect response to therapy? If we pre-identify rapid decliners from stable subjects, does this variable affect the response to whatever therapy is applied?
4. Can genetic analysis, genomics, proteomics, microbial and other biomarkers in the blood and cheeks provide insight into the polymorphisms and other elements related to the etiology and pathology of the lung damage?

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting to University of Virginia ILD or Pulmonary clinic
* Family members accompanying patients (as control subjects)

Exclusion Criteria:

* Control subjects cannot have ILD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients receiving care in the UVA ILD or Pulmonary clinic
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2018-08-28 (Actual); Primary Completion 2035-08-31 (Estimated); Study Completion 2035-08-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Course of Disease | Yearly from date of consent until subject is lost to follow-up or death occurs, whichever comes first, assessed up to 144 months
  Course of disease in patients with ILD will be reviewed prospectively for the duration of the study
Subject deaths | Yearly from date of consent until subject is lost to follow-up or death occurs, whichever comes first, assessed up to 144 months
  Causes of death in patients with ILD will be reviewed prospectively for the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Imre Noth, MD, Principal Investigator — University of Virginia Health System; Yousef Althulth, MD, Study Director — University of Virginia Health System
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Coded and de-identified data and specimens will be shared with collaborators. MTAs and DUAs are in place for such collaborations. This study also includes a data security plan that includes protective measures for sharing of data between investigators.